CLINICAL TRIAL: NCT03405077
Title: Harnessing Technology for Training Clinicians to Deliver Interpersonal Psychotherapy
Brief Title: Interpersonal Psychotherapy Online Training Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201408037
Record Dates: First submitted 2017-12-12; First posted 2018-01-19 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Eating Disorder
Keywords: interpersonal psychotherapy; treatment; training; dissemination and implementation; eating disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPT Online Training (Experimental): Therapists in this study will be trained in IPT using an online platform. The program is self-paced but will have a deadline; the suggested pace is at least 12 hours spaced over 2 months. The guided online training program was developed in collaboration with 3C institute, an award-winning research and development company that creates web- and evidence-based programs. Content will be adapted from "gold-standard" training.
  Interventions: Behavioral: IPT Online Training

INTERVENTIONS:
Behavioral: IPT Online Training — First, college mental health clinicians will complete baseline online questionnaires and deliver their usual treatment to 1 or 2 clients with symptoms of eating disorders. Then, they will complete the guided online training program and post-training assessments. Next, they will treat 1 or 2 different clients with eating disorders and complete post-training assessments. As part of the baseline and post-training assessments, clinicians will complete a telephone-based simulation assessment with staff raters, in which the investigators will recreate a client session and rate how well the clinicians adhere to IPT in treating the simulated client. The guided on-line training program will ultimately be compared to the "gold standard" training.

SUMMARY:
Interpersonal psychotherapy (IPT) is an evidence-based therapy for the treatment of eating disorders (including binge eating disorder, bulimia nervosa, and disordered eating not meeting full diagnostic criteria). On a basic level, IPT is a time-limited treatment that helps the client understand the relationship between symptoms and social interactions. Traditional training methods require substantial cost, time, and resources, making evidence-based treatments difficult to disseminate. As such, college clinicians are not typically trained in IPT delivery, which prevents their clients from reaping the potential benefits of treatment. This study will attempt to show how technology can overcome such barriers to training dissemination.

The purpose of this study is to see if online training in IPT is as effective as in-person training. To find out, the following procedures will occur: First, college mental health clinicians will complete baseline online questionnaires and deliver their usual treatment to 1 or 2 clients with symptoms of eating disorders. Then, they will complete the guided online training program and post-training assessments. Next, they will treat 1 or 2 different clients with eating disorders and complete post-training assessments. As part of the baseline and post-training assessments, clinicians will complete a telephone-based simulation assessment with staff raters, in which the investigators will recreate a client session and rate how well the clinicians adhere to IPT in treating the simulated client. The guided on-line training program will ultimately be compared to the "gold standard" training (the group receiving in-person training in an associated, IRB-approved study, # 201111113).

ELIGIBILITY:
THERAPISTS:

Inclusion criteria:

* Therapist must be a staff member at the counseling center and have a patient case-load large enough to be able to complete data collection at the different time points (>8 hours/week)
* Staff member is expected to continue working at the counseling center for several years • Postdocs who anticipate to be at their center for at least one year are eligible

Exclusion criteria:

* Therapists from all universities affiliated with the NIH-funded trial (IRB# 201111113)
* Therapists working less than 8 hours/week
* Therapists who are anticipating leaving employment at the recruited counseling center within the time frame of the study including, but not limited to trainees and interns
* Therapists for whom their administrative duties preclude seeing a sufficient number of clients to be able to complete data collection at the different study time points
* Therapists who do not see students seeking treatment for eating disorders
* Individuals who are non-degreed trainees (i.e., psychology interns)

STUDENTS:

Inclusion criteria:

* Student patients of therapists who seek counseling services at their respective schools
* Students exhibiting symptoms of an eating disorder

Exclusion criteria:

• Students exhibiting symptoms of anorexia nervosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Treatment fidelity: Adherence | 1-3 years
  Therapist's adherence to the procedures of IPT. This will be assessed using the IPT Fidelity Assessment. This scale was developed for the current study and was informed by work done by the Veterans' Health Administration, previous work conducted by the Principal Investigators of the current trial, and by other IPT researchers training therapists to conduct evidence-based treatments.

SECONDARY OUTCOMES:
Treatment fidelity: Competence | 1-3 years
  Therapist's level of competence in applying the procedures of IPT. This will be assessed using the IPT Fidelity Assessment. This scale was developed for the current study and was informed by work done by the Veterans' Health Administration, previous work conducted by the Principal Investigators of the current trial, and by other IPT researchers training therapists to conduct evidence-based treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Wilfley, PhD, Principal Investigator — Scott Rudolph University Professor of Psychiatry, Medicine, Pediatrics, and Psychological & Brain Sciences, Washington University School of Medicine; Terry Wilson, PhD, Study Director — Oscar K. Buros Professor of Psychology, Rutgers University; Stewart Agras, MD, Study Director — Professor of Psychiatry (Emeritus), Stanford University, School of Medicine

IPD SHARING:
Plan to Share IPD: No